CLINICAL TRIAL: NCT00602381
Title: A Single Dose, Three-Treatment, Three-Period, Six-Sequence Crossover Bioequivalency Study of 450 mg Lithium Carbonate Extended Release Tablets Under Fasting Conditions
Brief Title: Bioequivalency Study of 450 mg Lithium Carbonate Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, Drug Regulatory Affairs and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LITH-08
Record Dates: First submitted 2007-09-19; First posted 2008-01-28 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lithium

SUMMARY:
The objective of this study was to assess the bioequivalence of two Roxane lithium carbonate 450 mg extended release tablet formulations compared to GlaxoSmithKline's Eskalith CR 450 mg extended release tablet under fasting conditions using a single-dose, randomized, three-treatment, three-period, six-sequence crossover design.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

* Participation in a clinicl trial within 30 days prior to study initiation.
* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2002-11; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Baseline, Three period, Fourteen day washout

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Herron, MD, Principal Investigator — Arkansas Research
Locations (1):
- Arkansas Research, Little Rock, Arkansas, United States